CLINICAL TRIAL: NCT04674462
Title: Understanding Poor Vaccine Responses to Hepatitis B Vaccination
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-01782
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CpG-adjuvanted HBV Vaccine (Experimental)
  Interventions: Biological: CpG-adjuvanted HBV Vaccine
- Traditional HBV Vaccine (Active Comparator)
  Interventions: Biological: Traditional HBV Vaccine

INTERVENTIONS:
Biological: CpG-adjuvanted HBV Vaccine — Subjects receiving CpG-adjuvanted HBV vaccine will require two doses at 0 and 1 month after initiation. The second dose will be considered the same as the one month time point following the first dose.
  Arms: CpG-adjuvanted HBV Vaccine
Biological: Traditional HBV Vaccine — Subjects receiving traditional HBV vaccine series will require three doses at 0, 1, and 6 months after initiation. The second dose will be considered the same as the one month time point following the first dose.
  Arms: Traditional HBV Vaccine

SUMMARY:
Vaccines have prevented countless infections but poor vaccine responses remain a major challenge in many scenarios. Hepatitis B vaccine nonresponses are common but immunologically not well-understood.

This study aims to study the immunology of hepatitis B vaccine responses by comparing traditional HBV vaccine, which is associated with nonresponses in some patients, to CpG-adjuvanted HBV vaccine, which is associated with far fewer rates of nonresponses. This research will build upon prior studies of the human immune response to infection to gain a deeper understanding of the complexity of these responses. This information will be broadly useful as many vaccine candidates fail due to lack of immunogenicity, potentially enabling improved vaccine design and better protection.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Must be able to understand and sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. Known chronic HBV infection
2. Pregnancy
3. Known clinically significant anemia or contraindication to phlebotomy; i.e., anti-coagulation therapy or clinically significant thrombocytopenia
4. Any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study
5. Use of immune-suppressing medications in the 30 days prior to enrollment HIV/AIDS patients will be included in the study as these patients often have poor responses to HBV vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Weak Vaccine Response | Month 1 Post-Final Dose
  Weak vaccine response is defined as Hepatitis B surface antigen antibodies <= 10 mIU/mL (i.e. plasma anti-Hepatitis B surface antibody titer that is undetectable or below the cuff)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Herati, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to ramin.herati@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT04674462/ICF_000.pdf